CLINICAL TRIAL: NCT03857165
Title: A Multicenter, Randomized, Double-blind, Placebo Controlled, Dose Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of SAP-001 in Gout Patients With Hyperuricemia
Brief Title: Placebo Controlled, Dose Escalation Study to Evaluate Safety, Pharmacokinetics & Efficacy of SAP-001 in Gout Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanton Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Shanton Pharma Pte. Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAP-001; SAP001-1-001 (Other: SHANTON PHARMA CO., LTD.)
Record Dates: First submitted 2018-10-18; First posted 2019-02-27 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2019-11

CONDITIONS: Gout, Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Intervention Model Description: Single ascending dose with placebo control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose SAP-001 (Experimental): SAP-001 (Experimental drug) low dose versus placebo
  Interventions: Drug: SAP-001
- Mid dose SAP-001 (Experimental): SAP-001 (Experimental drug) mid dose versus placebo
  Interventions: Drug: SAP-001
- High dose SAP-001 (Experimental): SAP-001 (Experimental drug) high dose versus placebo
  Interventions: Drug: SAP-001

INTERVENTIONS:
Drug: SAP-001 — SAP-001 or placebo treatment in a 3:1 randomization ratio.

SUMMARY:
This is a Phase I, Multicenter, Randomized, Double-blind, Placebo controlled, Dose-escalation study to evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of SAP-001 in Gout Patients with Hyperuricemia. The study will be single dose ascending cohorts across three doses with a placebo control arm.

DETAILED DESCRIPTION:
A total of 24 eligible adult subjects will be randomized in a 3:1 randomization ratio into two blinded treatment groups in the three dose cohorts with matching placebo arm. The duration of the observation would be 5 days for each subject with a single SAP-001 dosing to evaluate safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and efficacy of oral SAP-001 (once daily) in adults gout patients with hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between 18 and 75 years of age, inclusive.
2. Body mass index (BMI) between 19 and 42 kg/m^2 at screening, inclusive.
3. Serum uric acid (sUA) levels ≥7.5 mg/dL at screening.
4. Patients must meet all the American College of Rheumatology scoring criteria for the classification of primary gout (Neogi et al., 2015).
5. Patients who are not taking any UA-lowering medications 1 month prior to the dose of study drug.
6. Is a nonsmoker or light smoker (smokes fewer than 10 cigarettes per day).
7. Female patients cannot be pregnant or lactating/breast-feeding and will either be postmenopausal (female patients who state they are postmenopausal should have had cessation of menses for>1 year and have serum follicle stimulating hormone [FSH] levels >40 mIU/mL and serum estradiol < 20 pg/mL or a negative estrogen test), surgically sterile (including bilateral tubal ligation, salpingectomy [with or without oophorectomy], surgical hysterectomy, or bilateral oophorectomy [with or without hysterectomy]) for at least 3 months prior to Screening, or will agree to use, from the time of Check-in (Day -1) until 90 days following the last dose of study drug, the following forms of contraception: double-barrier method, hormonal contraceptives, barrier with spermicide, diaphragm or cervical cap with spermicide, intrauterine device, oral, implantable, or injectable contraceptives, or a sterile sexual partner. All female patients will have a negative urine or serum pregnancy test result prior to enrollment in the study.
8. Male patients will either be surgically sterile or agree to use, from the time of Check-in (Day -1) until 90 days following the last dose of study drug, the following forms of contraception: male condom with spermicide and a female partner who is sterile or agrees to use hormonal contraceptives, female condom with spermicide, diaphragm or cervical cap with spermicide, intrauterine device, oral, implantable, or injectable contraceptives. Male patients will refrain from sperm donation from the time of Check-in (Day -1) until 90 days following the last dose of study drug.
9. Is capable of understanding the written informed consent, provides signed and witnessed written informed consent, and agrees to comply with protocol requirements.

Exclusion Criteria:

1. Has a history or presence of clinically significant (CS) cardiovascular, renal, pulmonary, hepatic, gallbladder or biliary tract, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease, which in the Investigator's opinion would not be suitable for the study.
2. Serum creatinine level > 1.5 mg/dL and/or estimated glomerular filtration (eGFR) by the Modification of Diet in Renal Disease (MDRD) rate ≤60 mL/min/1.73 m2 at screening. The MDRD formula is: GFR (mL/min/1.73 m2) = 175 × (Scr)-1.154 × (Age)-0.203 × (0.742 if female) × (1.212 if African American)
3. History of stomach or intestinal surgery (except that cholecystectomy, appendectomy, and/or hernia repair will be allowed).
4. History of prescription drug abuse, illicit drug use, or alcohol abuse according to medical history within 6 months prior to the Screening visit or any alcohol use for at least 48 hours prior to dosing on Day 1.
5. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C (HCV) antibody.
6. Clinically significant abnormal liver function test at screening or Check-in (Day -1), defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT)>1.5 times upper limit of normal (ULN) or total bilirubin >ULN; or a history of clinically significant acute or chronic hepatitis (including infectious, metabolic, autoimmune, genetic, ischemic, or other forms), hepatocirrhosis, or hepatic tumors.
7. Positive screen for alcohol or drugs of abuse (except for patients with a positive drug screen test if it is a result of a prescribed medication from their physician) at Screening and Check-in (Day -1).
8. History of a gout flare that is resolved within 14 days prior to first treatment with study drug (exclusive of chronic synovitis/arthritis).
9. Has a known hypersensitivity to URAT1 inhibitors, XOIs, or related compounds.
10. Receipt of any other investigational product within 30 days prior to the dose of study drug on Day 1or planning to take an investigational agent during the study.
11. Concomitant use of or treatment with any prescription drugs, herbal products, vitamins, minerals, and over-the-counter medications within 14 days prior to Check in (Day -1). Exceptions may be made on a case by case basis following discussion and agreement between the Investigator and the Sponsor.
12. Use of any drugs or nutrients known to modulate cytochrome P450 (CYP)3A activity or any strong or moderate inhibitors or inducers of CYP3A4, starting from 14 days prior to dose administration on Day 1 until the final end of study assessments, including but not limited to the following: inhibitors such as ketoconazole, miconazole, itraconazole, fluconazole, atazanavir, erythromycin, clarithromycin, ranitidine, cimetidine, verapamil, and diltiazem and inducers such as rifampicin, rifabutin, glucocorticoids, carbamazepine, phenytoin, phenobarbital, and St. John's wort.
13. Participated in strenuous exercise from 48 hours prior to Check-in (Day -1) or during the study through the final end of study assessment.
14. Has donated or lost a significant volume (>500 mL) of blood or plasma within 30 days prior to Check-in (Day -1).
15. Malignancy within 5 years of the screening visit.
16. Has problems understanding the protocol requirements, instructions, study related restrictions, and/or problems understanding the nature, scope, and potential consequences of participating in this clinical study.
17. Is unlikely to comply with the protocol requirements, instructions, and/or study related restrictions (e.g., uncooperative attitude, unavailable for follow up call, and/or improbability of completing the clinical study).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 5 days
  Safety and tolerability of single escalating dose SAP-001
Cmax | 5 days
  Maximum Plasma Concentration of SAP-001 in ng/mL
tmax | 5 days
  Time to maximum concentration in hours
AUC0-t | 5 days
  Area under the concentration-time curve from time 0 to time t, calculated using the linear trapezoidal rule for increasing values, and the log trapezoidal rule for decreasing values
AUC0-24h | 24 hours
  Area under the concentration-time curve from time 0 until 24 hours post dose, calculated using the linear trapezoidal rule for increasing values, and the log trapezoidal rule for decreasing values
λz | 5 days
  Apparent terminal elimination rate constant
t1/2 | 5 days
  Terminal elimination phase half-life of SAP-001, calculated as ln(2)/λz
CL/F | 5 days
  Total body clearance of SAP-001, calculated as Dose/AUC0-∞
Vz/F | 5 days
  Volume of distribution of SAP-001
MRT | 5 days
  Mean residence time in hours

SECONDARY OUTCOMES:
Serum uric acid (sUA) levels at various time points | 72 hours
  Serum uric acid (sUA) levels in mg/dL at various time points after oral administration of ascending single dose of SAP-001 or placebo
IL-1β | 24 hours
  Inflammatory cytokine IL-1β in pg/mL
IL-6 | 24 hours
  Inflammatory cytokine IL-6 in pg/mL
IL-8 | 24 hours
  Inflammatory cytokine IL-8 in pg/mL
TNFα | 24 hours
  Inflammatory cytokine TNFα in pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: John M Hill, MD, Principal Investigator — Accel Research Sites (Avail Clinical Research); Melanie Fein, Principal Investigator — High Point Clinical Trials Center; Peter Winkle, Principal Investigator — Anaheim Clinical Trials, LLC
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Avail - Accel Research Sites, DeLand, Florida
  - High Point Clinical Trials Center, High Point, North Carolina

IPD SHARING:
Plan to Share IPD: No